CLINICAL TRIAL: NCT06972004
Title: Preventing Loss of Independence Through Exercise in Community Living Centers: An Effectiveness-Implementation Trial
Brief Title: Preventing Loss of Independence Through Exercise in Community Living Centers
Acronym: PLIE-CLC
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: IIR 23-027; 23-027-02 (Other Grant/Funding Number: VA Health Systems Research); 1I01HX003817-01A2 (NIH)
Record Dates: First submitted 2025-05-06; First posted 2025-05-14 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Dementia; Cognitive Dysfunction
Keywords: health-related quality of life; Social Participation; Accidental Falls; Pain; Movement; Behavior; neurocognitive disorder; nursing homes; implementation science
MeSH Terms: conditions — Dementia; Cognitive Dysfunction; Pain; Behavior; Neurocognitive Disorders

STUDY DESIGN:
Intervention Model Description: The investigators propose to perform a hybrid type 2 effectiveness-implementation study with a stepped wedge cluster randomized trial (SW-CRT) design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PLIE-CLC (Other): Preventing Loss of Independence through Exercise (PLIÉ) is a multi-domain, mind-body, group movement program for people with dementia that improves quality of life. A stepped wedge cluster randomized trial design includes: 1) a baseline data collection phase where no clusters are exposed to the intervention; 2) sequential randomized crossover to the intervention (PLIÉ-CLC); and 3) analyses that account for time trends and correlations within clusters. Randomization of facilities to PLIÉ-CLC will simply delay rollout to sites randomized later in the sequence (like a wait-list control condition).
  Interventions: Behavioral: Preventing Loss of Independence through Exercise (PLIE)

INTERVENTIONS:
Behavioral: Preventing Loss of Independence through Exercise (PLIE) — Preventing Loss of Independence through Exercise (PLIÉ) is a multi-domain, mind-body, group movement program for people with dementia that improves quality of life.
  Classes begins and ends with fully body tapping/massaging and breathing exercises that bring participants into awareness of their bodies in the present moment and create a calming ritual. Participants are invited to share appreciations of things in their lives that make them feel happy or grateful. Instructors lead participants through progressive, functional movement sequences that are designed to be repetitive (to build procedural or "muscle" memory) and to build slowly in functional complexity over time. Movements are tailored to the ability levels of the group. Resting, breathing and mindful body awareness exercises are incorporated throughout each class to provide breaks and to improve focus and attention. A non-judgmental errorless learning process is used, and all movements are performed slowly and purposefully.
  Other Names: PLIE-CLC

SUMMARY:
Approximately 40,000 older Veterans who have complex care needs (for example, a combination of severe cognitive, physical, and mental health conditions) receive long-term care in VA Community Living Centers (CLCs). However, CLC staff members rarely receive specialized training in how to best engage and interact with these Veterans, which can lead to poor care quality, worsening of symptoms, staff burnout, and low morale throughout a facility. The investigators have developed a unique, mind-body, group movement program for Veterans with cognitive impairment called Preventing Loss of Independence through Exercise (PLIÉ) and found that it has physical, cognitive, social and emotional benefits in CLC residents. The investigators recently taught 50 staff members from a variety of professions in 5 CLCs to lead PLIÉ classes. The study will enable us to test whether the PLIÉ,LC staff training program improves outcomes for residents and to learn about the success and sustainment of the training.

DETAILED DESCRIPTION:
Background: Preventing Loss of Independence through Exercise (PLIÉ) is a unique, mind-body, group movement program for people living with cognitive impairment and dementia that has been found to have physical, cognitive, social, and emotional benefits. The investigators received a VA Innovators Award to implement PLIÉ in the San Francisco VA Community Living Center (CLC), where it became one of their most successful and popular programs. As part of the ongoing VA HSR&D pre-implementation grant (1I01 HX002764), the investigators have developed and piloted a remote PLIÉ staff training program and have successfully trained 50 interprofessional staff members at 5 CLCs. This study will enable us to test the effectiveness and implementation of PLIÉ-CLC.

Significance: VA CLCs serve approximately 40,000 Veterans annually, most of whom have one or more severe neurocognitive, mental health or physical impairments; yet CLC staff members typically do not receive specialized training in how to best engage and interact with these Veterans. This training and knowledge gap can result in poor care quality, declines in physical function, increased distressed behaviors, staff burnout, and low morale throughout a facility.

Innovation & Impact: PLIÉ-CLC provides an efficient format for delivering high-quality care to groups of residents with cognitive impairment. Veterans with complex care needs often receive care from different providers who do not necessarily communicate with each other about the residents' needs. PLIÉ-CLC provides a structured framework for interprofessional staff members to work together to simultaneously address residents' physical, social and mental health needs. In addition, PLIÉ-CLC provides an efficient experiential training model. Staff members, trainees and family members are invited to join classes where they can learn by doing and can directly observe the beneficial impact of the classes on residents.

Specific Aims: The goals of this study are to: 1) Determine the effectiveness of PLIÉ-CLC on resident, entered outcomes (primary outcome: physical function; secondary outcomes: social engagement, mood, cognitive function, behaviors, falls, and pain); 2) Determine the effectiveness of PLIÉ-CLC on person-centered care practices and organizational culture, including staff engagement, burnout, and workplace climate; 3) Evaluate implementation of PLIÉ-CLC, including reach, adoption, external facilitation, and fidelity; 4) Examine the extent to which PLIÉ-CLC is sustained after external facilitation support has ended.

Methodology: The investigators proposed to achieve these Specific Aims by performing a Type 2 Hybrid Effectiveness%2Implementation study using a stepped wedge cluster randomized trial design. This design will enable us to assess the effectiveness of PLIÉ-CLC at the resident (Aim 1) and organizational (Aim 2) levels and the implementation process itself at the clinician and organizational levels (Aims 3, 4). The investigators will use a concurrent mixed methods approach to qualitative and quantitative data collection and analysis guided by the Practical, Robust Implementation and Sustainability Model (PRISM).

Next Steps/Implementation: The investigators will work with study partners in the VA Office of Geriatrics and Extended Care, Office of Patient Centered Care & Cultural Transformation, and Mental Health & Suicide Prevention to use the findings from this effectiveness-implementation trial to inform decisions about sustainable roll out and implementation of PLIÉ-CLC nationwide.

ELIGIBILITY:
Inclusion Criteria:

CLC internal facilitators/champions Inclusion criteria:

* Full-time CLC clinical staff member (including registered nurses, certified nursing assistants, nurse aids, recreation therapists, occupational therapists, physical therapists, mental health professionals or others)
* Willingness to facilitate PLIÉ-CLC implementation at their site
* Willingness to participate in initial and debrief site visit

PLIÉ-CLC staff instructors Inclusion criteria:

* CLC clinical staff member or volunteer interested in learning to lead PLIÉ-CLC classes
* Willingness to participate in remote training process
* Willingness to lead PLIÉ classes locally, including tracking attendance and other process measures
* Willingness to participate in initial and debrief site visits and biweekly check-ins

Veteran residents of Community Living Centers (CLCs) Inclusion criteria:

* Long-stay resident (have resided at the facility for at least 45 days and are not expected to be discharged during the study period)
* Not planning to be discharged within the next 12 months
* Not receiving hospice care.
* Cognitive impairment
* Ability to sit in a standard chair or wheelchair unaided for a 1-hour class
* English language fluency

CLC directors Inclusion criteria:

* Recommended by VHA leader as likely to be 'early adopter' based on successful implementation of program such as STAR-VA OR
* g based on patient population (primarily palliative care or long stay maintenance/custodial care

Exclusion Criteria:

CLC internal facilitators/champions exclusion Criteria:

- Planning to leave the facility in next 12 months

PLIÉ-CLC staff instructors exclusion criteria:

- Planning to leave the facility in next 12 months

Veteran residents of Community Living Centers (CLCs) exclusion Criteria:

* Comatose
* Bedbound
* Severe hearing, visual or communication challenges (i.e., unable to hear, see or understand well enough to participate)
* Limited life expectancy (e.g., eligible for hospice)
* Lack of ability to consent/assent to study procedures

CLC Directors exclusion criteria:

- Lack of willingness or interest in participating

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 288 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2028-11-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
MDS Section G (Resident Physical Function) | -6 to 0 months (baseline), 0-6 months, 9 months, 2 months
  The investigators will assess change in resident physical function using the Minimum Data Set (MDS) 3.0. The MDS has nearly 400 data elements, including cognitive function, physical functioning, behavioral symptoms, mood symptoms, pain and falls. Facility MDS coordinators (typically RNs) complete assessments for all Veterans in CLCs on admission, quarterly, and with changes in status. Reliability of the MDS is "very good" to "excellent" on most data items and scales. The investigators are using an 17-item MDS physical function measure that combines items from sections G1 (assistance needed with bed mobility, transferring, walking in room, walking in facility, and locomotion) and G3 (balance in standing, walking, turning around, getting on and off the toilet, and transferring) to create a continuous score that ranges from 0 (fully independent and steady at all times) to 136 (unable to do with or without assistance).

SECONDARY OUTCOMES:
RISE (Staff) | -6 to 0 months (baseline), 0-6 months, 9 months, 12 months
  The Revised Index of Social Engagement (RISE) proxy will be completed by CLC staff at 0, 6, and 12 months and includes 6 yes/no questions about Veteran engagement (e.g., Is the Veteran at ease interacting with others).
MDS (Behavior) | -6 to 0 months (baseline), 0-6 months, 9 month, 12 months
  The investigators will assess change in resident behavior using the Minimum Data Set (MDS) 3.0.
MDS (Cognition) | -6 to 0 months (baseline), 0-6 months, 9 months, 12 months
  The investigators will assess change in resident cognition using the Minimum Data Set (MDS) 3.0.
MDS (Mood) | -6 to 0 months (baseline), 0-6 months, 9 months, 12 months
  The investigators will assess change in resident mood using the Minimum Data Set (MDS) 3.0.
MDS (Pain) | -6 to 0 months (baseline), 0-6 months, 9 months, 12 months
  The investigators will assess change in resident pain using the Minimum Data Set (MDS) 3.0.
MDS (Falls) | -6 to 0 months (baseline), 0-6 months, 9 months, 12 months
  The investigators will assess change in resident falls using the Minimum Data Set (MDS) 3.0.
PLIE Experience Scale for Staff | 0-6 months, 9 months, 12 months
  Staff and residents reported survey after intervention. PLIÉ Experience measure at the end of the implementation period (6 months) and again 6 months later (12 months). This measure includes 6 items with parallel versions for staff and residents as well as an overall rating. In addition, the survey includes open-ended questions about what participants enjoyed most, changes noticed in themselves and others, and suggestions for improvements.
PLIE Clinical Note | 0-6 months, 9 months, 12 months
  PLIÉ clinical note free-text descriptions from a 15% random sample of residents per site will be used to assess staff observation and documented change over time across resident secondary outcomes domains.
PC-PAL (Staff) | -6 to 0 months (baseline), 0-6 months, 9 months, 12 months
  The Staff Person-Centered Care Practices in Assisted Living (PC-PAL) measure [is a validated tool to assess the degree to which the culture and practices of long-term care settings promote person-centered care in the following areas: workplace practices, social connectedness, individualized care and practices, atmosphere, and caregiver-resident relationships. To measure the impact of PLIE-CLC on key person-centered care domains among staff participants, the investigators will ask staff to complete 12 items from PC-PAL at 0, 6 and 12 months.
AES (Staff) | -6 to 0 months (baseline), 0-6, 9, 12 months
  The VA All Employee Survey (AES) includes validated questions related to organizational culture and employee engagement. Most items are rated on a 5-point Likert scale (strongly disagree to strongly agree). The investigators will ask staff participants to complete three subscales: workplace performance (6 items); job satisfaction (3 items); and burnout (3 items) at 0, 6 and 12 months.
Reach | 1-6, 9, 12 months
  The investigators will use CDW data to assess the proportion and characteristics (e.g., gender, race/ethnicity) of eligible residents engaged in PLIÉ-CLC beyond initial training cases at (6, 9 and 12 months).
Qualitative Interviews | 2, 4, 6, 12 months
  Qualitative semi-structured data will be collected from staff regarding the following topics: Blended facilitation & Training effectiveness, facilitation & training experience, leadership and organizational support.
NoMAD - Survey | 0, 6, 12 months
  Staff surveys include the 25-item Normalization Measurement Development (NoMAD). Scores on this validated measure are used to identify patterns across NPT domains, e.g., if the intervention makes sense to CLC staff (coherence) but is failing due to low engagement (cognitive participation).
Adoption | 3-6, 9, 12 months
  Adoption will be measured by the total number and proportion of trained staff at each site who deliver PLIÉ groups after the training program. Data will be obtained from VA corporate data .
Clinical Sustainability Assessment Tool (CSAT) | 0, 6, 12 months
  Sustainment capacity, or the ability to maintain PLIE-CLC and its benefits over time, will be evaluated with the 35-item Clinical Sustainability Assessment Tool (CSAT). Internal facilitations/champions and staff will rate the CSAT independently over time (0, 6, 12 months) to track progress and inform sustainment planning.
Staff level fidelity to PLIE Protocol | 5, 6, 9, 12 months
  The investigators will assess staff fidelity to the PLIÉ-CLC protocol and through staff teaching practicum assessments and chart review of at least a 10% random sample of PLIÉ-CLC clinical notes, which include checkboxes of key PLIÉ principles taught as well as free text descriptions of resident response. The investigators will assess for variations at the staff and facility levels.
PLIE Class Experience for Residents | 6, 12 months
  Staff and residents reported survey after intervention. PLIÉ Experience measure at the end of the implementation period (6 months) and again 6 months later (12 months). This measure includes 6 items with parallel versions for staff and residents as well as an overall rating. In addition, the survey includes open-ended questions about what participants enjoyed most, changes noticed in themselves and others, and suggestions for improvements

CONTACTS AND LOCATIONS:
Overall Officials: Francesca M Nicosia, PhD MA, Principal Investigator — San Francisco VA Medical Center, San Francisco, CA; Linda L. Chao, PhD BS, Principal Investigator — San Francisco VA Medical Center, San Francisco, CA
Locations (1):
- San Francisco VA Medical Center, San Francisco, CA, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No